CLINICAL TRIAL: NCT00949104
Title: A Study to Assess the Role of Oral Sucrose in Reducing the Pain to Orogastric Tube Insertion in Preterm Neonates
Brief Title: Role of Oral Sucrose in Reducing the Pain to Orogastric Tube Insertion in Preterm Neonates
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: DR Vikram Datta, Lady Hardinge Medical College,New Delhi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OGTPAIN
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Pain in Preterm Neonates
Keywords: Sucrose; pain; neonate; preterm; orogastric tube
MeSH Terms: conditions — Pain; Premature Birth | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sucrose (Active Comparator): 1 ml of 24% sucrose was administered 2 minutes before the procedure
  Interventions: Drug: Sucrose
- Placebo (Placebo Comparator): Double distilled water
  Interventions: Drug: Double distilled water

INTERVENTIONS:
Drug: Sucrose — 1 ml of 24% sucrose was administered 2 minutes prior to the procedure
  Other Names: 24%Sucrose
  Arms: Sucrose
Drug: Double distilled water — 1 ml of double distilled water (Placebo) was administered 2 minutes prior to the procedure
  Arms: Placebo

SUMMARY:
RESEARCH HYPOTHESIS Orally administered sucrose 2 minutes prior to the procedure of OGT insertion reduces pain associated with the procedure.

AIMS AND OBJECTIVES:

To study the effect of 24% oral sucrose on decreasing the painful response to orogastric tube insertion .

DETAILED DESCRIPTION:
MATERIAL & METHODS

PARTICPANTS:

INCLUSION CRITERIA: The enrolled participants must fulfill the following inclusion criteria:

* All pre-terms ( < 37 weeks of gestational age.)
* Within the first 7 days postnatal days (</=168 hours).
* Clinically stable from respiratory, hemodynamic and metabolic point of view.
* Who have not received any painful stimulus at least 30 minutes prior to the intervention.
* Requiring routine orogastric tube insertion within the first 7 days of life.
* Only the first attempt at putting OGT in controlled NICU environment will be considered

EXCLUSION CRITERIA: The neonates with the following characteristics will be excluded from the study:

* Neonates requiring ventilatory support.
* Neonates requiring oxygen supplementation.
* Having any facial congenital anomalies.
* Having any neurological impairment.
* Receiving opiates or born to mothers receiving opiates.
* New born babies to whom muscle relaxants, sedatives and analgesics have been administered.
* With grade 3 and 4 IVH.
* With major congenital anomalies
* Any history of birth trauma especially involving face or scalp (including cephalhematoma/ subgaleal bleed).
* Face presentation.

INTERVENTIONS:

There will be two groups in the study ( group A & group B). The enrolled neonates will be administered either a sterile solution of 24% sucrose or double distilled water orally. These solutions will be prepared under all sterile precautions by the laboratory staff unrelated to the study, and packed in 2 ml sterile syringes further covered with opaque sealed envelopes bearing serially numbered patient codes. The composition of these packets would be decided by a senior consultant in the department of pharmacology who would have the access to the randomization sequence and would be uninvolved in the present study. Fresh solutions will be prepared daily and unused solutions will be discarded at the end of the day to be replaced with identically numbered solutions from the laboratory. All study solutions will be stored in the refrigerator at 2-8 0C until they are used.

The patients will be enrolled into the study only after an informed written consent has been obtained from either of the parent/ caregiver. 2 minutes prior to procedure, 1 ml of the solution marked with patients's serial number will be administered orally to the patient by a nurse using the syringe. The procedure would involve putting a 5-6 Fr. OGT in the neonate which will be done by a group of 8-10 nurses who have been specially trained in this procedure. This insertion of OGT will be done 2 min post administration of test solution by a nurse who will be blinded to the contents of the solution.

The whole procedure (beginning 2 minutes before the OGT insertion and continuing till 4 minutes after it is inserted) will be video recorded on a fixed camera focusing on the face of the patient. Neonate will be monitored using a non invasive vital signs monitor to monitor his heart rate and SpO2 changes during the entire procedure and for 2 minutes post procedure. The highest heart rate and lowest SpO2 obtained during the procedure till 2 minutes post procedure will be recorded. The research candidate will evaluate the pain response to the procedure according to the PIPP scale at time t=pre-procedure, t=intra-procedure,t=post 30 sec, t=post 1min, & t=post 2 min; wherein t denotes the time at which tube is inserted into the oral cavity. The research candidate will also monitor the time taken in the OGT insertion using a stopwatch. The neonatal nurse putting the OGT will rate the procedure as easy, difficult or very difficult.

OUTCOMES:

PRIMARY OUTCOME: Painful response, as assessed by the PIPP scale. SECONDARY OUTCOME: Maximum heart rate and minimum oxygen saturation recorded during the procedure.

SAMPLE SIZE CALCULATION:The sample size was calculated based on the assumption that there would be a decrease of at least 20% in the pain scores in the study population with the intervention and using a alpha error of 0.05 and a power of 90% the sample size was calculated to be 55 each in both the groups ie a total of 110 neonates.

RANDOMISATION:Block Randomisation using computer generated random sequences with a block size of 4 each.

SEQUENCE GENERATION:

Block randomization using computer generated random sequences will be used.

ALLOCATION CONCEALMENT:

This will be done by the pharmacy who will pack the sucrose and the double distilled water (control/placebo) into identical containers and opaque sealed envelopes sequentially labeled according to randomization code.

IMPLEMENTATION:

Randomization sequence will be generated by a senior consultant in the department of pharmacology .The participants will be enrolled for the study by the candidate according to the serial number as the candidate will be blinded.

BLINDING:

The participants, the research candidate,the nursing staff administering the intervention as well as the investigators assessing the painful response will be blinded to the group assignment

STATISTICAL METHODS: Descriptive statistics will be calculated.Between groups comparison of continuous variables will be done with the help of t test for parametric data and by Mann Whitney test for non parametric data.The proportion and frequencies will be calculated using the chi square test.

ELIGIBILITY:
Inclusion Criteria:

* All pre-terms ( < 37 weeks of gestational age.)
* Within the first 7 days postnatal days (</=168 hours).
* Clinically stable from respiratory, hemodynamic and metabolic point of view.
* Who have not received any painful stimulus at least 30 minutes prior to the intervention.
* Requiring routine orogastric tube insertion within the first 7 days of life.
* Only the first attempt at putting OGT in controlled NICU environment will be considered

Exclusion Criteria:

The neonates with the following characteristics will be excluded from the study:

* Neonates requiring ventilatory support.
* Neonates requiring oxygen supplementation.
* Having any facial congenital anomalies.
* Having any neurological impairment.
* Receiving opiates or born to mothers receiving opiates.
* New born babies to whom muscle relaxants, sedatives and analgesics have been administered.
* With grade 3 and 4 IVH.
* With major congenital anomalies
* Any history of birth trauma especially involving face or scalp (including cephalhematoma/ subgaleal bleed).
* Face presentation.

Ages: 1 Hour to 167 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Painful response as assessed by PIPP Scale | Pre procedure,Intra procedure,post 30 sec,post 1 min,post 2 minutes

SECONDARY OUTCOMES:
Maximum heart rate and minimum oxygen saturation | pre procedure,intra procedure,post 30 seconds,post 1 minute,post 2 minute

CONTACTS AND LOCATIONS:
Overall Officials: VIKRAM DATTA, MD,DNB, Study Chair — LADY HARDINGE MEDICAL COLLEGE,NEW DELHI,INDIA
Locations (1):
- Lady Hardinge Medical College, New Delhi, New Delhi, India

REFERENCES:
- [Derived] Pandey M, Datta V, Rehan HS. Role of sucrose in reducing painful response to orogastric tube insertion in preterm neonates. Indian J Pediatr. 2013 Jun;80(6):476-82. doi: 10.1007/s12098-012-0924-4. Epub 2012 Dec 21. PMID 23263970